CLINICAL TRIAL: NCT01438424
Title: A Preliminary Assessment of Safety and Antiviral Activity of Open-label Entecavir in Subjects With Chronic Hepatitis B Following Monotherapy in Other Entecavir Trials
Brief Title: Safety and Antiviral Activity of Entecavir in Participants With Chronic Hepatitis B Following Monotherapy in Other Entecavir Trials
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI463-901
Record Dates: First submitted 2011-09-16; First posted 2011-09-22 (Estimated); Results first posted 2012-08-23 (Estimated); Last update posted 2012-08-23 (Estimated); Status verified 2012-07

CONDITIONS: Hepatitis B Virus; HBV
MeSH Terms: conditions — Hepatitis B | interventions — entecavir; Lamivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Entecavir, 1.0 mg, with or without lamivudine (Experimental)
  Interventions: Drug: Entecavir; Drug: Lamivudine

INTERVENTIONS:
Drug: Entecavir — Tablets, Oral, 1.0 mg, once daily
  Other Names: Baraclude
Drug: Lamivudine — Oral, 100 mg, daily

SUMMARY:
The purpose of this study is to provide entecavir to participants who have completed another entecavir trial without achieving virologic response or who relapsed during postdosing follow-up.

ELIGIBILITY:
Key inclusion criteria:

* Age of 16 years and older
* Receipt of entecavir or lamivudine in a previous entecavir study.

Participants who were, based on their response to entecavir:

* Virologic nonresponders at Week 48
* Partial virologic responders who became nonresponders during the second year of treatment
* Partial virologic responders at Week 96
* Complete responders who relapsed during postdosing follow-up

  * Decompensated liver disease in AI463-048 that met 1 or more of the following criteria:
* Nonresponse to adefovir after at least 24 weeks of treatment
* Partial response to adefovir after 96 weeks of treatment
* Complete response to adefovir after relapsing during postdosing follow-up
* Demonstrated intolerance to adefovir

  * Except for those participants enrolled from AI463-048, compensated liver disease.

Key exclusion criteria:

* HIV coinfection
* Receiving nephrotoxic or hepatotoxic agents
* Ongoing opportunistic infections
* Hemoglobin level <11.0 g/dL except for those enrolled from AI463-048
* Platelet count <70,000 mm^3 except for those enrolled from AI463-048
* Absolute granulocyte count <1,500 cells/mm^3
* Recent history of pancreatitis (within 24 weeks prior to first dose of therapy)
* Current evidence of ascites requiring paracentesis, hepatic encephalopathy, or variceal bleeding, except for those enrolled from AI463-048
* Known history of allergy to nucleoside analogues.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1053 (Actual)
Dates: Start 2001-01; Primary Completion 2009-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb

REFERENCES:
- [Derived] Manns MP, Akarca US, Chang TT, Sievert W, Yoon SK, Tsai N, Min A, Pangerl A, Beebe S, Yu M, Wongcharatrawee S. Long-term safety and tolerability of entecavir in patients with chronic hepatitis B in the rollover study ETV-901. Expert Opin Drug Saf. 2012 May;11(3):361-8. doi: 10.1517/14740338.2012.653340. Epub 2012 Jan 11. PMID 22233350

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 1053 participants enrolled, 1051 received treatment.
Groups:
- Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine: Participants originally received 0.5 mg of entecavir once daily (QD) with lamivudine, but protocol later amended to 1.0 mg of entecavir QD without lamivudine.
Period: Overall Study
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Started | 1051 (Received treatment)
Completed | 634 (Completed treatment)
Not Completed | 417
Not completed — Continuing treatment | 29
Not completed — Minimal virologic response | 95
Not completed — Not identified | 55
Not completed — Withdrawal by Subject | 104
Not completed — Progression of chronic hepatitis B | 22
Not completed — Death | 22
Not completed — Adverse Event | 17
Not completed — Lost to Follow-up | 17
Not completed — Abnormal laboratory test result | 14
Not completed — Need for drug prohibited by protocol | 14
Not completed — Pregnancy | 7
Not completed — No longer met inclusion criteria | 1
Not completed — Participant noncompliance | 20

BASELINE CHARACTERISTICS:
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Age, Customized [Median (Standard Deviation); unit: Years] | 41 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 241
  Male | 810
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian/Pacific Islander | 544
  White | 481
  Black/African American | 18
  Missing | 2
  Native Hawaiian/Other Pacific Islander | 2
  Other | 2
  Filipino | 1
  Hispanic/Latino | 1
Region: Continent [Number; unit: Participants]
  Asia | 451
  Europe | 334
  North America | 141
  South America | 125
Age [Mean (Full Range); unit: Years] | 41 [17 to 78]

OUTCOME MEASURES:

1. Secondary Outcome: Overall Study: Percentage of Participants With Sustained HBV DNA Level <300 Copies/mL by PCR Assay
Time Frame: Study entry to Week 192
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Groups:
- Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine: Participants originally received 0.5 mg of entecavir QD with lamivudine, but protocol later amended to 1.0 mg of entecavir QD without lamivudine.
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Percentage of participants
  At study entry (n=1051) | 17
  Week 48 (n=905) | 63
  Week 96 (n=691) | 67
  Week 144 (n=597) | 73
  Week 192 (n=485) | 78

2. Secondary Outcome: Overall Study: Percentage of Participants With Sustained HBV DNA <10^4 Copies/mL by PCR Assay
Time Frame: Study entry to Week 192
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Percentage of participants
  At study entry (n=1051) | 28
  Week 48 (n=905) | 76
  Week 96 (n=691) | 77
  Week 144 (n=597) | 81
  Week 192 (n=485) | 85

3. Secondary Outcome: Overall Study: Percentage of Participants by HBV DNA Category by PCR Assay
Description: Observed values.
Time Frame: Baseline to Week 192
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Groups:
- Entecavir, 1.0 mg, With or Without Lamivudine: Participants received 1 mg of entecavir QD with or without lamivudine.
Arm/Group | Entecavir, 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Percentage of participants
  Baseline: <300 copies/mL (n=1051) | 17 (4)
  Baseline: 300 - <1.0E3 copies/mL (n=1051) | 4 (8)
  Baseline: 1.0E3 - <1.0E4 copies/mL (n=1051) | 8 (13)
  Baseline: 1.0E4 - <1.0E5 copies/mL (n=1051) | 8 (11)
  Baseline: 1.0E5 - <1.0E6 copies/mL (n=1051) | 12
  Baseline: 1.0E6 - <1.0E7 copies/mL (n=1051) | 13
  Baseline: 1.0E7 - <1.0E8 copies/mL (n=1051) | 8
  Baseline: 1.0E8 - <1.0E9 copies/mL (n=1051) | 11
  Baseline: 1.0E9 - <1.0E10 copies/mL (n=1051) | 13
  Baseline: >= 1.0E10 copies/mL (n=1051) | 6
  Week 192: < 300 copies/mL (n=485) | 78
  Week 192: 300 - <1.0E3 copies/mL (n=485) | 3
  Week 192: 1.0E3 - <1.0E4 copies/mL (n=485) | 3
  Week 192: 1.0E4 - <1.0E5 copies/mL (n=485) | 4
  Week 192: 1.0E5 - <1.0E6 copies/mL (n=485) | 2
  Week 192: 1.0E6 - <1.0E7 copies/mL (n=485) | 2
  Week 192: 1.0E7 - <1.0E8 copies/mL (n=485) | 1
  Week 192: 1.0E8 - <1.0E9 copies/mL (n=485) | 5
  Week 192: 1.0E9 - <1.0E10 copies/mL (n=485) | 2
  Week 192: >= 1.0E10 copies/mL (n=485) | 0

4. Primary Outcome: Overall Study: Number of Participants With Death As Outcome, Any Adverse Event (AE), Grade 3-4 AEs, Serious Adverse Events (SAEs), and Discontinuations Due to AEs
Description: An AE is a new unfavorable symptom, sign, or disease or worsening of a preexisting condition that may not be causally related to treatment. An SAE is an unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling. ALT=alanine transaminase; ULN=upper limit of normal.
Time Frame: Continuously from Day 1 through Week 240
Population: All participants who received at least 1 dose of study drug in the current study.
Measure: Number; unit: Participants
Groups:
- Entecavir, 0.5 or 1.0 mg QD, With or Without Lamivudine: Participants originally received 0.5 mg of entecavir once daily (QD) with lamivudine, but protocol later amended to 1.0 mg of entecavir QD without lamivudine. All participants, regardless of dosing or regimen, included in these safety analyses.
Arm/Group | Entecavir, 0.5 or 1.0 mg QD, With or Without Lamivudine
Number analyzed (Participants) | 1051
Participants
  Deaths on treatment | 18
  Deaths off treatment | 9
  SAEs on treatment | 169
  Discontinuations due to AEs on treatment | 14
  Any AE on treatment | 900
  Grade 3 and 4 AEs on treatment | 203
  Malignancies on and off treatment | 35
  ALT flares (ALT>2*entry and >10*ULN) on treatment | 32
  Hepatic disease progression on and off treatment | 33

5. Secondary Outcome: Overall Study: Mean HBV DNA Level by PCR Assay
Time Frame: Study entry to Week 216
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Mean (Standard Deviation); unit: log10 copies/mL
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
log10 copies/mL
  At study entry (n=1051) | 6.14 (2.667)
  Week 12 (n=1017) | 3.87 (1.749)
  Week 24 (n=1010) | 3.62 (1.684)
  Week 48 (n=905) | 3.37 (1.543)
  Week 72 (n=769) | 3.31 (1.549)
  Week 96 (n=691) | 3.34 (1.592)
  Week 120 (n=629) | 3.32 (1.665)
  Week 144 (n=597) | 3.34 (1.826)
  Week 168 (n=514) | 3.18 (1.663)
  Week 192 (n=485) | 3.19 (1.757)
  Week 216 (n=455) | 3.20 (1.789)

6. Secondary Outcome: Overall Study: Percentage of Participants Who Achieved a Loss of Hepatitis B e Antigen (HBeAg)
Description: Observed values.
Time Frame: Study entry to Week 216
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Percentage of participants
  At study entry (n=1051) | 34
  Week 12 (n=935) | 40
  Week 24 (n=939) | 42
  Week 48 (n=864) | 46
  Week 72 (n=752) | 45
  Week 96 (n=679) | 50
  Week 120 (n=609) | 51
  Week 144 (n=587) | 53
  Week 168 (n=518) | 58
  Week 192 (n=491) | 60
  Week 216 (n=436) | 59

7. Secondary Outcome: Overall Study: Percentage of Participants With HBeAg Seroconversion
Description: Observed values. Seroconversion=negative HBeAg with detectable anti-HBe antibody.
Time Frame: Study entry to Week 216
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Percentage of participants
  At study entry (n=1051) | 30
  Week 12 (n=931) | 33
  Week 24 (n=934) | 34
  Week 48 (n=862) | 36
  Week 72 (n=755) | 32
  Week 96 (n=678) | 34
  Week 120 (n=607) | 36
  Week 144 (n=587) | 37
  Week 168 (n=517) | 39
  Week 192 (n=491) | 42
  Week 216 (n=434) | 40

8. Secondary Outcome: Overall Study: Mean Alanine Transaminase (ALT) Levels
Description: Observed values.
Time Frame: Study entry to Week 216
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Entecavir, 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
U/L
  At study entry (n=1051) | 109.4 (170.5)
  Week 12 (n=1049) | 48.77 (48.68)
  Week 24 (n=1029) | 42.10 (36.83)
  Week 48 (n=942) | 37.06 (34.20)
  Week 72 (n=835) | 38.10 (41.90)
  Week 96 (n=740) | 39.30 (46.35)
  Week 120 (n=675) | 37.43 (28.97)
  Week 144 (n=627) | 38.51 (38.95)
  Week 168 (n=563) | 36.80 (29.06)
  Week 192 (n=528) | 37.36 (30.44)
  Week 216 (n=482) | 38.43 (55.09)

9. Secondary Outcome: Overall Study: Percentage of Participants Who Achieved ALT Normalization
Description: ULN=upper limit of normal. ALT normalization=ALT levels ≤1.0*ULN.
Time Frame: Study entry to Week 216
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Percentage of participants
  At study entry (n=1019) | 40
  Week 48 (n=942) | 75
  Week 144 (n=627) | 74
  Week 216 (n=482) | 78

10. Secondary Outcome: Week 192: Percentage of Participants With Histologic Improvement (Efficacy Evaluable Cohort)
Description: The Knodell Histologic Activity Index scores stage of necrosis and grade of inflammation in liver biopsies. Components are necrosis near the portal vein, intralobular degeneration and focal necrosis, portal inflammation, and fibrosis. The 4 components are scored from 1 to 4 and 1 to 10 (necrosis near the portal vein) and combined for a total score, with 22 being the highest possible score. Higher the score for each component=greater liver damage. Histologic improvement=a ≥2-point reduction in total Knodell score and no worsening in fibrosis. Cohort participants had to have adequate baseline and long-term biopsy samples and baseline Knodell necroinflammatory scores ≥2.
Time Frame: Baseline to Week 192
Population: Subset of participants who who had evaluable paired liver biopsy results at Phase 3 study baseline and on their last observed biopsies performed in the current study. (n=number of evaluable participants)
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 57
Percentage of participants
  Histologic improvement (n=56) (Week 48) | 73 [60 to 84]
  Histologic improvement (n=57) (Long-term biopsy) | 96 [88 to 100]

11. Secondary Outcome: Week 192: Percentage of Participants With Improvement in Fibrosis (Efficacy Evaluable Cohort)
Description: The Ishak Modification for Hepatic Activity Index (HAI) scores necroinflammatory activity in chronic hepatitis. 0=no fibrosis, 1=fibrosis expansion of some portal areas, 2=fibrosis expansion of most portal areas, 3=fibrosis expansion of most portal areas with occasional bridging, 4=fibrosis expansion of portal areas with marked bridging, 5=incomplete cirrhosis, 6=probable or definite cirrhosis. Higher score=more severe necrosis. Improvement in fibrosis=≥1-point reduction in HAI score. Cohort participants had to have adequate baseline and long-term biopsy samples and baseline Knodell scores ≥2.
Time Frame: Baseline to Week 192
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 57
Percentage of participants
  Improvement in fibrosis (n=56) (Week 48) | 32 [20 to 46]
  Improvement in fibrosis (n=57) (Long-term biopsy) | 88 [76 to 95]

12. Primary Outcome: Overall Study: Number of Participants With Normal Hematology Values at Baseline and Abnormalities in Hematology Laboratory Test Results Through Week 240
Description: Hemoglobin (g/dL): Grade (Gr) 1=9.5-11.0; Gr 2=8.0-<9.5; Gr 3=6.5-<8.0; Gr 4=<6.5 White blood cells (cells/mm^3): Gr 1=2,500-<4,000; Gr 2=1,000-<2,500; Gr 3=800-<1,000; Gr 4=<800. Neutrophils (cells/mm^3): Gr 1=1000-<1500; Gr 2=750-<1000; Gr 3=500-<750; Gr 4=<500. Platelets (cells/mm^3): Gr 1=75,000-99,000; Gr 2=50,000-<75,000; Gr 3=20,000-<50,000; Gr 4=<20,000. Prothrombin time (seconds): Gr 1=1.01-<1.26*ULN; Gr 2=1.26-<1.51 *ULN; Gr 3=1.51-3*ULN; Gr 4=>3*ULN. INR: Gr 1=1.24-1.5; Gr 2=1.5-2; Gr 3=2-3; Gr 4=>3. INR=international normalized ratio; ULN=upper limit of normal. .
Time Frame: Day 1 of treatment through Week 240
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Participants
  Hemoglobin (All grades) (n=1007) | 49
  White blood cells (All grades) (n=950) | 226
  Neutrophils (All grades) (n=1002) | 109
  Platelets (All grades) (n=979) | 51
  Protrombin time (All grades) (n=746) | 226
  INR (All grades)(n=746) | 214
  Hemoglobin (Grades 3-4) (n=1007) | 2
  White blood cells (Grades 3-4) (n=950) | 1
  Neutrophils (Grades 3-4) (n=1002) | 21
  Platelets (Grades 3-4) (n=979) | 1
  Prothrombin time (Grades 3-4) (n=746) | 21
  INR (Grades 3-4) (n=746) | 12

13. Primary Outcome: Overall Study: Number of Participants With Normal Pancreatic Enzyme and Renal Function Values at Baseline and Abnormalities in Pancreatic Enzyme and Renal Function Laboratory Test Results at End of Dosing
Description: Amylase: Grade 1=1.10-<1.40*ULN; Grade 2=1.40-< 2.10*ULN; Grade 3=2.10-5.00*ULN; Grade 4=>5.00*ULN. Lipase: Grade 1.1-<1.4*ULN; Grade 2=1.4-<2.1*ULN; Grade 3=2.1-5.0*ULN; Grade 4=>5.0*ULN. Creatinine: Grade 1=1.10-< 1.60*ULN; Grade 2=1.60-<3.10*ULN; Grade 3=3.10-6.00*ULN; Grade 4=>6.00*ULN. Blood urea nitrogen (BUN): Grade 1=1.25-<2.60*ULN; Grade 2=2.60-<5.10*ULN; Grade 3=5.10-10*ULN; Grade 4=>10*ULN. ULN=upper limit of normal.
Time Frame: Day 1 of treatment through Week 240
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Participants
  Amylase (All grades) (n=875) | 179
  Lipase (All grades) (n=390) | 126
  Amylase (Grades 3-4) (n=875) | 13
  Lipase (Grades 3-4) (n=390) | 38
  BUN/Urea (All grades) (n=998) | 57
  Creatinine (All grades) (n=1000) | 61
  BUN/Urea (Grades 3-4) (n=998) | 0
  Creatinine (Grades 3-4) (n=1000) | 2

14. Primary Outcome: Overall Study: Number of Participants With Normal Electrolyte and Fasting Glucose Values at Baseline and Abnormalities in Electrolyte and Fasting Glucose Laboratory Test Results at End of Dosing
Description: Hypochloremia: Grade (Gr) 1=90-93; Gr 2=85-<90; Gr 3=80-<85; Gr 4=40-<80. Hyperchloremia: Gr 1=113-<117; Gr 2=117-<121; Gr 3=121-125; Gr 4>125. Hypocarbia: Gr 1=19-21; Gr 2=15-<19; Gr 3=41-45; Gr 4=>45. Hypercarbia: Gr 1=31-36; Gr 2=37-40; Gr 3=41-45; Gr 4=>45. Hyponatremia: Gr 1=130-132; Gr 2=123-<130; Gr 3=116-<123; Gr 4<116. Hypernatremia: Gr 1=148-<151; Gr 2=151-<158; Gr 3=158-165; Gr 4=>165. Hypokalemia: Gr 1=3-3.4; Gr 2=2.5-<3; Gr 3=2-<2.5; Gr 4=<2. Hyperkalemia: Gr 1=5.6-<6.1; G2=6.1-<6.6; Gr 3=6.6-7; Gr 4=>7. Hypoglycemia: Gr 1=55-64; Gr 2=40-<55; Gr 3=30-< 40; G4=-<30. Hyperglycemia: Gr 1=116-<161; Gr 2=161-<251; Gr 3=251-500; Gr 4>500.
Time Frame: Day 1 of treatment through Week 240
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Participants
  Hypochloremia (mEq/L) (All grades) (n=982) | 44
  Hyperchloremia (mEq/L) (All grades) (n=982) | 76
  Hypocarbia (mEq/L) (All grades) (n=831) | 285
  Hypercarbia (mEq/L) (All grades) (n=831) | 148
  Hyponatremia (mEq/L) (All grades) (n=1003) | 68
  Hypernatremia (mEq/L) (All grades) (n=1003) | 106
  Hypokalemia (mEq/L) (All grades) (n=993) | 135
  Hyperkalemia (mEq/L) (All grades (n=993) | 42
  Hypochloremia (mEq/L) (Grades 3-4) (n=982) | 3
  Hyperchloremia (mEq/L) (Grades 3-4) (n=982) | 7
  Hypocarbia (mEq/L) (Grades 3-4) (n=831) | 14
  Hypercarbia (mEq/L) (Grades 3-4) (n=831) | 2
  Hyponatremia (mEq/L)(Grades 3-4) (n=1003) | 2
  Hypernatremia (mEq/L) (Grades 3-4) (n=1003) | 5
  Hypokalemia (mEq/L) (Grades 3-4) (n=993) | 1
  Hyperkalemia (mEq/L) (Grades 3-4) (n=993) | 6
  Hypoglycemia (mg/dL) (All grades) (n=521) | 47
  Hyperglycemia (mg/dL) (All grades) (n=521) | 150
  Hypoglycemia (mg/dL) (Grades 3-4) (n=521) | 3
  Hyperglycemia (mg/dL) (Grades 3-4) (n=521) | 4

15. Secondary Outcome: Overall Study: Percentage of Participants With a Confirmed ≥1 log10 Increase From Nadir in HBV DNA by PCR Assay
Time Frame: Baseline to Week 144
Population: Participants who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 1051
Percentage of participants | 18

16. Primary Outcome: Week 144: Number of Participants With Death As Outcome, Any AE, Grade 3-4 AEs, SAEs, Discontinuations Due to AEs, and Abnormalities in Selected Laboratory Test Results
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling. AST=aspartate aminotransferase; ULN=upper limit of normal.
Time Frame: Continuously from Day 1 through Week 144
Population: Participants enrolled up to Week 144 who received at least 1 dose of study drug in the current study. (n=number of evaluable participants)
Measure: Number; unit: Participants
Groups:
- Entecavir, 0.5 or 1.0 mg QD, With or Without Lamivudine: Participants originally received 0.5 mg of entecavir QD with lamivudine, but protocol later amended to 1.0 mg of entecavir QD without lamivudine. All participants, regardless of dosing or regimen, included in these safety analyses.
Arm/Group | Entecavir, 0.5 or 1.0 mg QD, With or Without Lamivudine
Number analyzed (Participants) | 996
Participants
  Deaths on study | 13
  Malignant neoplasms | 17
  SAEs | 107
  Discontinuations due to AEs | 13
  Any AE | 842
  Grade 3 and 4 AEs | 156
  ALT flares (ALT>2*entry and >10*ULN) | 29
  ALT >5.0*ULN | 93
  AST >5.0*ULN | 53
  Total bilirubin >2.5*ULN | 22
  Lipase >2.0*ULN | 71
  Creatinine ≥0.5 mg/dL from baseline | 6
  Hypocarbia | 4

17. Secondary Outcome: Percentage of Participants Who Achieved HBV DNA <300 Copies/mL by PCR Assay, Loss of HBeAG, Seroconversion, and ALT ≤1.0*Upper Limit of Normal (ULN) (Entecavir Continuous Treatment Cohort)
Description: The Entecavir Continuous Treatment Cohort consisted of participants from study AI463-022 (NCT00035633) who were nucleoside-naive HBeAg-positive and enrolled in the current study with ≤35 days off treatment between the last dose in AI463-022 and the first dose in the current. This cohort is considered to be on continuous entecavir treatment and permitted assessment of continuous administration of entecavir in AI463-022 and the current study.
Time Frame: Baseline to Weeks 48, 96, 144, 192, and 240
Population: Participants enrolled from study AI463-022 who were nucleoside-naive, HBeAg-positive and enrolled in the current study with ≤35 days off treatment between the last dose in AI463-022 and the first dose in the current study and were evaluable. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 146
Percentage of participants
  Week 48: HBV DNA <300 copies/mL (n=146) | 55
  Week 96: HBV DNA <300 copies/mL (n=140) | 83
  Week 144: HBV DNA <10^4 copies/mL (n=131) | 89
  Week 192: HBV DNA < 10^4 copies/mL (n=108) | 91
  Week 240: HBV DNA <300 copies/mL (n=94) | 94
  Week 48: Loss of HBeAg (n=146) | 1
  Week 96: Loss of HBeAg (n=140) | 4
  Week 144: Loss of HBeAg (n=132) | 30
  Week 192: Loss of HBeAg (n=111) | 39
  Week 240: Loss of HBeAg (n=95) | 41
  Week 48: Seroconversion (n=146) | 1
  Week 96: Seroconversion (n=140) | 3
  Week 144: Seroconversion (n=133) | 17
  Week 192: Seroconversion (n=111) | 16
  Week 240: Seroconversion (n=95) | 17
  Week 48: ALT ≤1.0*ULN (n=146) | 65
  Week 96: ALT ≤1.0*ULN (n=140) | 78
  Week 144: ALT ≤1.0*ULN (n=134) | 77
  Week 192: ALT ≤1.0*ULN (n=112) | 86
  Week 240: ALT ≤1.0*ULN (n=98) | 80

18. Secondary Outcome: Percentage of Participants Who Achieved HBV DNA <300 and <10^4 Copies/mL by PCR Assay and ALT ≤1.0*Upper Limit of Normal (ULN) (Entecavir Retreatment Cohort)
Description: The Entecavir Retreatment Cohort consisted of participants who were nucleoside-naive, HBeAg-negative and enrolled from BMS study AI463-027 with >60 days off treatment between the last dose in AI463-027 and the first dose in the current study. This cohort permitted assessment of entecavir, 1.0 mg, provided as retreatment in the current study.
Time Frame: Baseline to Weeks 48, 96, and 144
Population: Participants enrolled from study AI463-027 who were nucleoside-naive, HBeAg-negative and had >60 days off treatment between the last dose in AI463-027 and the first dose in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 99
Percentage of participants
  Week 48: HBV DNA <300 copies/mL (n=119) | 88
  Week 48: HBV DNA <10^4 copies/mL (n=88) | 87
  Week: 48: ALT ≤1.0*ULN (n=95) | 83
  Week 96: HBV DNA <300 copies/mL (n=74) | 91
  Week: 96: ALT ≤1.0*ULN (n=76) | 79
  Week 144: HBV DNA <300 copies/mL (n=57) | 95
  Week 144: ALT ≤1.0*ULN (n=66) | 86

19. Secondary Outcome: Week 96: Percentage of Participants Who Achieved HBV DNA <300 Copies/mL by PCR Assay, Loss of HBeAg, HBeAg Seroconversion, and ALT ≤1.0*ULN (Lamivudine Continuous Switch Cohort)
Description: The Lamivudine Continuous Switch Cohort consisted of participants who were nucleoside-naive, HBeAg-positive and received lamivudine in BMS study AI463-022 (NCT00035633) and enrolled in the current study with ≤35 days off treatment between end of dosing in AI463-022 and the switch to entecavir in the current study. This cohort permitted assessment of entecavir, 1.0 mg, provided as switch therapy in the current study.
Time Frame: Baseline to Week 96
Population: Participants enrolled from AI463-022 who received lamivudine, were nucleoside-naive HBeAg-positive, and had ≤35 days off treatment between end of dosing in AI463-022 and the switch to entecavir in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 183
Percentage of participants
  HBV DNA <300 copies/mL (n=147) | 58
  Achieved loss of HbeAg (n=129) | 25
  Achieved HBeAg seroconversion (n=129) | 8
  Achieved ALT ≤1.0*ULN (n=154) | 76

20. Secondary Outcome: Week 144: Percentage of Participants Who Achieved HBV DNA <300 Copies/mL by PCR Assay and ALT ≤1.0*ULN (Lamivudine Continuous Switch Cohort)
Description: as for outcome 19
Time Frame: Baseline to Week 144
Population: as for outcome 19
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 183
Percentage of participants
  HBV DNA <300 copies/mL (n=130) | 65
  Achieved ALT ≤1.0*ULN (n=135) | 68

21. Primary Outcome: Week 192: Number of Participants With Death As Outcome, Any AE, Grade 3-4 AEs, SAEs, Discontinuations Due to AEs, and Abnormalities in Selected Laboratory Test Results
Description: An AE is any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not necessarily have a causal relationship with treatment. An SAE is any unfavorable medical event that at any dose results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; or requires or prolongs hospitalization. CTC Grade 1=mild; Grade 2=moderate; Grade 3=severe; Grade 4=life-threatening or disabling. ALT=alanine aminotransferase; ULN=upper limit of normal.
Time Frame: Continuously from Day 1 through Week 192
Population: Participants who enrolled from Phase 3 studies of nucleoside-naive HBeAg-positive (AI463-022) and HBeAg-negative (AI463-027) participants and received at least 1 dose of study drug in the current study up to Week 192. (n=number of evaluable participants)
Measure: Number; unit: Participants
Arm/Group | Entecavir, 0.5 or 1.0 mg QD, With or Without Lamivudine
Number analyzed (Participants) | 1006
Participants
  Deaths on study | 18
  Malignant neoplasms | 27
  SAEs | 135
  Discontinuations due to AEs | 11
  Any AE | 862
  Grade 3 and 4 AEs | 174
  ALT flares (ALT>2*entry and >10*ULN) | 30
  ALT >5.0*ULN | 175
  Total bilirubin >2.5*ULN | 32
  Lipase >2.0*ULN | 81
  Creatinine ≥0.3 mg/dL from baseline | 80
  Hypocarbia Grades 3-4 | 5

22. Secondary Outcome: Week 96: Percentage of Participants Who Achieved HBV DNA <300 Copies/mL by PCR Assay and ALT ≤1.0*ULN (Lamivudine Retreatment Switch Cohort)
Description: The Lamivudine Retreatment Switch Cohort consisted of participants who were nucleoside-naive HBeAg negative and enrolled from BMS study AI463-027 (NCT00035789) with >60 days between end of dosing in AI463-027 and the switch to entecavir in the current study. This cohort permitted assessment of entecavir, 1.0 mg, provided as switch therapy in the current study.
Time Frame: Baseline to Week 96
Population: Participants enrolled from AI463-027 who were nucleoside-naive HBeAg-negative, received lamivudine, and had >60 days between end of dosing in AI463-027 and the switch to entecavir in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 123
Percentage of participants
  HBV DNA <300 copies/mL (n=69) | 97
  ALT ≤1.0*ULN (n=81) | 81

23. Secondary Outcome: Week 144: Percentage of Participants Who Achieved HBV DNA <300 Copies/mL by PCR Assay and ALT ≤1.0*ULN (Lamivudine Retreatment Switch Cohort)
Description: as for outcome 22
Time Frame: Baseline to Week 144
Population: Participants enrolled from study AI463-027 who were nucleoside-naive HBeAg-negative and had >60 days off treatment between the last dose in AI463-027 and the first dose in the current study. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 123
Percentage of participants
  HBV DNA <300 copies/mL (n=67) | 99
  Achieved ALT ≤1.0*ULN (n=73) | 85

24. Primary Outcome: Off-treatment Follow-up: Percentage of Participants With Sustained Hepatitis B Virus (HBV) DNA <10,000 Copies by Polymerase Chain Reaction (PCR) Assay (Amendment 11 Cohort)
Description: The Amendment 11 Cohort consisted of participants who were hepatitis B e antigen (HBeAg) negative and who had compensated liver disease, a minimum of 192 weeks (4 years) of treatment with entecavir, HBV DNA <300 copies/mL by PCR assay for ≥48 weeks before end of dosing and on the last observed result ≤24 weeks prior to end of dosing, and serum ALT levels ≤1.0*ULN at the end of study drug dosing.ALT=alanine aminotransferase; ULN=upper limit of normal.
Time Frame: End of dosing to Week 48 off-treatment follow-up
Population: Participants who were HBeAg negative and who had compensated liver disease, a minimum of 192 weeks (4 years) of treatment with entecavir, HBV DNA <300 copies/mL by PCR assay for ≥48 weeks before end of dosing and on the last observed result ≤24 weeks prior to end of dosing, and serum ALT levels ≤1.0*ULN at the end of study drug dosing.
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 29
Percentage of participants
  End of dosing current study | 100
  Off-treatment Week 48 | 21

25. Secondary Outcome: Off-treatment Follow-up: Percentage of Participants With Sustained HBV DNA <1,000, <300, and <10,000 Copies/mL by PCR Assay and With ALT ≤1*ULN (Amendment 11 Cohort)
Description: The Amendment 11 Cohort consisted of participants who were HBeAg negative and who had compensated liver disease, a minimum of 192 weeks (4 years) of treatment with entecavir, HBV DNA <300 copies/mL by PCR Assay for ≥48 weeks before end of dosing and on the last observed result ≤24 weeks prior to end of dosing, and serum ALT levels ≤1.0*ULN at the end of study drug dosing. ULN=upper limit of normal.
Time Frame: End of dosing to Weeks 48 and 96 off-treatment follow-up
Population: Participants who were HBeAg negative and who had liver disease, a minimum of 192 weeks of entecavir treatment, HBV DNA <300 copies/mL by PCR assay for ≥48 weeks before end of dosing and on the last observed result ≤24 weeks before end of dosing, and serum ALT levels ≤1.0*ULN at the end of study drug dosing. (n=number of evaluable participants)
Measure: Number; unit: Percentage of participants
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 29
Percentage of participants
  Off-treatment Week 48 <1000 copies/mL | 10
  Off-treatment Week 96 <1000 copies/mL | 10
  Off-treatment Week 48 <300 copies/mL | 7
  Off-treatment Week 96 <300 copies/mL | 3
  Off treatment Week 96 <10,000 copies/mL | 14
  Off treatment Week 48: ALT ≤1*ULN | 31
  Off treatment Week 96: ALT ≤1*ULN | 24

26. Secondary Outcome: Off-treatment Follow-up: Mean Change in HBV DNA (Amendment 11 Cohort)
Description: The Amendment 11 Cohort consisted of participants who were HBeAg negative and who had compensated liver disease, a minimum of 192 weeks (4 years) of treatment with entecavir, HBV DNA <300 copies/mL by PCR assay for ≥48 weeks before end of dosing and on the last observed result ≤24 weeks prior to end of dosing, and serum ALT levels ≤1.0*ULN at the end of study drug dosing.
Time Frame: End of dosing to Weeks 48 and 96 off-treatment follow-up
Population: Participants who were HBeAg negative and who had liver disease, a minimum of 192 weeks of entecavir treatment, HBV DNA <300 copies/mL by PCR assay for ≥48 weeks before end of dosing and on the last observed result ≤24 weeks before end of dosing, and had serum ALT levels ≤1.0*ULN at the end of study drug dosing. (n=number of evaluable participants)
Measure: Mean (Standard Error); unit: Log10 copies/mL
Arm/Group | Entecavir, 0.5 or 1.0 mg, With or Without Lamivudine
Number analyzed (Participants) | 29
Log10 copies/mL
  Off-treatment Week 48 | 1.54 (0.336)
  Off-treatment Week 96 | 1.18 (0.326)

ADVERSE EVENTS:
Groups:
- Adefovir, 10 mg: Participants who received adefovir concomitantly at postdosing follow-up
- Entecavir, 0.02588 mg; Entecavir, 0.1 mg; Entecavir, 1.0 mg: Participants originally received lower doses of entecavir QD with lamivudine, but protocol later amended to 1.0 mg of entecavir QD without lamivudine.
- Entecavir, 0.5 mg: Participants received entecavir QD with lamovidine
- Lamovidine, 100 mg: Participants originally received lamovidine with entecavir
- Missing: Category missing
- Placebo: Participants originally assigned to placebo before protocol change to study drug.
Arm/Group | Adefovir, 10 mg | Entecavir, 0.02588 mg | Entecavir, 0.1 mg | Entecavir, 0.5 mg | Entecavir, 1.0 mg | Lamovidine, 100 mg | Missing | Placebo
Serious Adverse Events (participants affected / at risk) | 7/35 | 0/1 | 3/29 | 57/336 | 15/123 | 87/523 | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 27/35 | 0/1 | 25/29 | 274/336 | 94/123 | 439/523 | 2/2 | 1/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir, 10 mg (N=35) | Entecavir, 0.02588 mg (N=1) | Entecavir, 0.1 mg (N=29) | Entecavir, 0.5 mg (N=336) | Entecavir, 1.0 mg (N=123) | Lamovidine, 100 mg (N=523) | Missing (N=2) | Placebo (N=2)
VESTIBULAR NEURONITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ASCITES (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LUNG NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CELLULITIS (Infections and infestations) | 1 | 0 | 0 | 2 | 0 | 1 | 0 | 0
DEVICE RELATED INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
VASCULAR ENCEPHALOPATHY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
NEPHROLITHIASIS (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
OBSTRUCTIVE UROPATHY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HAEMORRHAGIC FEVER (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MALFORMATION VENOUS (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VERTIGO POSITIONAL (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
INGUINAL HERNIA (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0
HEPATIC HAEMATOMA (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PERITONITIS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MYOLIPOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PANCREATIC CARCINOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
SPINAL COLUMN INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CHOLECYSTITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
CHRONIC HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEPATIC NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 6 | 3 | 16 | 0 | 0
TRANSAMINASES INCREASED (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
TUBERCULIN TEST POSITIVE (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BENIGN BREAST NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
AMOEBIASIS (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
BILIARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HEPATITIS B (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OSTEOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MEDICATION ERROR (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SIALOADENITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
STREPTOCOCCAL SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
SUBCUTANEOUS ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BURN OESOPHAGEAL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 6 | 0 | 0
APPENDICITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 0
HAEMOLYTIC ANAEMIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MANIA (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
HEPATITIS INFECTIOUS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PYELONEPHRITIS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VENTRICULAR EXTRASYSTOLES (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
MACULAR OEDEMA (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
URINARY INCONTINENCE (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OVARIAN CYST (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
EYE PENETRATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYPERTENSION (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HUMERUS FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SPINAL CORD INJURY CERVICAL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
HEPATIC NEOPLASM MALIGNANT RECURRENT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BLOOD AMYLASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LIPASE INCREASED (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SJOGREN'S SYNDROME (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
ARRHYTHMIA (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
POLYNEUROPATHY (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
KLEBSIELLA SEPSIS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
URETHRAL DISORDER (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ELECTRICAL BURN (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
FALL (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEAD INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OESOPHAGEAL VARICES HAEMORRHAGE (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
INFLAMMATION (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
MULTIPLE MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
LIVER DISORDER (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CEREBRAL HAEMATOMA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
UTERINE POLYP (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ANAL FISTULA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
FOOD POISONING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
GASTRIC VARICES HAEMORRHAGE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
LYMPHOPROLIFERATIVE DISORDER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
SPINAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OBESITY (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
CHONDROPATHY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
EPILEPSY (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
INTRACRANIAL HAEMATOMA (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ANAL ABSCESS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0
CHRONIC SINUSITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DENGUE FEVER (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
AUTOIMMUNE THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
COMPLETED SUICIDE (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CALCULUS URETERIC (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ADRENAL MASS (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
PULMONARY MASS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
TONSILLAR DISORDER (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ELECTIVE SURGERY (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
HAEMATOMA (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
GENITAL INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
TRANSITIONAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
PYREXIA (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
JAUNDICE (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
HAEMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SOFT TISSUE INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
TYPHOID FEVER (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEPATIC NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 4 | 0 | 8 | 0 | 0
LYMPHOMA CUTIS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
MALIGNANT PERITONEAL NEOPLASM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
METASTASES TO BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
LABORATORY TEST ABNORMAL (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ADENOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
BILE DUCT CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CEREBRAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HYDRONEPHROSIS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DIPLOPIA (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
FEMORAL NECK FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
OESOPHAGEAL ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
VOMITING (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEPATIC FAILURE (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
GASTRIC CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
INVESTIGATION (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HEADACHE (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
IIIRD NERVE PARESIS (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PARAESTHESIA (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
LIVER ABSCESS (Infections and infestations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
PERITONSILLAR ABSCESS (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PNEUMONIA (Infections and infestations) | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0
CORONARY ARTERY STENOSIS (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
SKIN NEOPLASM EXCISION (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
SQUAMOUS CELL CARCINOMA OF SKIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
PAIN (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
JOINT INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OVERDOSE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0
HEPATITIS (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
COLON CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
VIRAL INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HAEMATEMESIS (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
INTERVERTEBRAL DISC DEGENERATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
CEREBRAL HAEMORRHAGE (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
DIZZINESS (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
DIARRHOEA INFECTIOUS (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
EAR INFECTION (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
NEPHROPATHY (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
OVARIAN CYST RUPTURED (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VARICES OESOPHAGEAL (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
VARICOSE VEIN (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
ABSCESS (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adefovir, 10 mg (N=35) | Entecavir, 0.02588 mg (N=1) | Entecavir, 0.1 mg (N=29) | Entecavir, 0.5 mg (N=336) | Entecavir, 1.0 mg (N=123) | Lamovidine, 100 mg (N=523) | Missing (N=2) | Placebo (N=2)
HEPATIC ENCEPHALOPATHY (Nervous system disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 0 | 0 | 23 | 5 | 52 | 0 | 0
ASCITES (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 0 | 2 | 0 | 0
DUODENAL ULCER (Gastrointestinal disorders) | 3 | 0 | 0 | 6 | 0 | 5 | 0 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 2 | 0 | 0 | 16 | 2 | 14 | 0 | 0
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 15 | 4 | 31 | 0 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 2 | 0 | 0 | 5 | 2 | 6 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 2 | 0 | 4 | 12 | 2 | 37 | 1 | 0
ASTHENIA (General disorders) | 2 | 0 | 1 | 13 | 4 | 25 | 0 | 0
FATIGUE (General disorders) | 2 | 0 | 7 | 36 | 13 | 63 | 0 | 0
GALLBLADDER POLYP (Hepatobiliary disorders) | 2 | 0 | 1 | 9 | 1 | 13 | 0 | 0
HEPATIC STEATOSIS (Hepatobiliary disorders) | 0 | 0 | 2 | 14 | 8 | 21 | 0 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 9 | 0 | 5 | 89 | 27 | 154 | 0 | 0
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 6 | 33 | 11 | 86 | 0 | 0
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 5 | 35 | 5 | 59 | 0 | 0
LIPODYSTROPHY ACQUIRED (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
HYPERTENSION (Vascular disorders) | 1 | 0 | 4 | 44 | 13 | 63 | 0 | 0
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3 | 13 | 7 | 36 | 0 | 0
RESTLESS LEGS SYNDROME (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
HAEMATURIA (Renal and urinary disorders) | 1 | 0 | 1 | 21 | 4 | 29 | 0 | 0
DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 | 1 | 4 | 1 | 0
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 2 | 3 | 1 | 14 | 0 | 0
NASOPHARYNGITIS (Infections and infestations) | 8 | 0 | 5 | 60 | 18 | 83 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 0 | 5 | 22 | 9 | 44 | 0 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0 | 5 | 46 | 12 | 84 | 0 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 2 | 2 | 0 | 3 | 0 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 7 | 2 | 7 | 0 | 0
TACHYCARDIA (Cardiac disorders) | 0 | 0 | 0 | 3 | 0 | 3 | 1 | 0
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 | 0 | 7 | 42 | 7 | 67 | 0 | 0
DERMATITIS CONTACT (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 1 | 3 | 0 | 0
TOOTHACHE (Gastrointestinal disorders) | 2 | 0 | 1 | 16 | 4 | 38 | 0 | 0
INFLUENZA LIKE ILLNESS (General disorders) | 0 | 0 | 1 | 10 | 3 | 18 | 1 | 0
OEDEMA PERIPHERAL (General disorders) | 2 | 0 | 0 | 1 | 1 | 13 | 0 | 0
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0 | 0 | 18 | 3 | 29 | 1 | 0
LACERATION (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 4 | 3 | 7 | 0 | 0
INSOMNIA (Psychiatric disorders) | 2 | 0 | 4 | 26 | 6 | 49 | 0 | 0
UPPER RESPIRATORY TRACT CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 1 | 0 | 1 | 0 | 0
PALPITATIONS (Cardiac disorders) | 0 | 0 | 2 | 9 | 0 | 12 | 0 | 0
DYSPEPSIA (Gastrointestinal disorders) | 3 | 0 | 8 | 25 | 10 | 44 | 1 | 0
FOOD POISONING (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0
PYREXIA (General disorders) | 7 | 0 | 7 | 38 | 10 | 43 | 0 | 0
PROSTATITIS (Reproductive system and breast disorders) | 0 | 0 | 2 | 1 | 0 | 3 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 4 | 48 | 15 | 77 | 0 | 0
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 5 | 2 | 7 | 0 | 0
CONJUNCTIVITIS (Eye disorders) | 1 | 0 | 0 | 8 | 1 | 5 | 1 | 0
DIARRHOEA (Gastrointestinal disorders) | 5 | 0 | 1 | 44 | 12 | 69 | 1 | 0
MALAISE (General disorders) | 2 | 0 | 2 | 5 | 1 | 20 | 0 | 0
MUSCLE RUPTURE (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
RASH (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 11 | 7 | 14 | 0 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 5 | 12 | 2 | 26 | 0 | 0
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 7 | 2 | 20 | 0 | 0
HEADACHE (Nervous system disorders) | 3 | 0 | 13 | 69 | 16 | 131 | 1 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 28 | 7 | 37 | 1 | 0
PAIN (General disorders) | 0 | 0 | 2 | 2 | 1 | 11 | 0 | 0
SEASONAL ALLERGY (Immune system disorders) | 0 | 0 | 1 | 7 | 3 | 19 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 2 | 17 | 4 | 20 | 0 | 0
INFLUENZA (Infections and infestations) | 4 | 0 | 4 | 45 | 13 | 53 | 1 | 0
RHINITIS (Infections and infestations) | 0 | 0 | 0 | 11 | 3 | 15 | 1 | 0
TONSILLITIS (Infections and infestations) | 2 | 0 | 1 | 11 | 1 | 11 | 0 | 0
ECZEMA (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 8 | 3 | 11 | 0 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 16 | 5 | 13 | 0 | 0
DIZZINESS (Nervous system disorders) | 2 | 0 | 2 | 24 | 5 | 44 | 1 | 0
HAEMORRHOIDS (Gastrointestinal disorders) | 3 | 0 | 0 | 6 | 2 | 14 | 0 | 0
CHEST PAIN (General disorders) | 2 | 0 | 3 | 8 | 6 | 20 | 0 | 0
HYPERSENSITIVITY (Immune system disorders) | 2 | 0 | 0 | 1 | 0 | 11 | 0 | 0
HERPES ZOSTER (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 7 | 0 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 | 0 | 3 | 16 | 4 | 31 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.